CLINICAL TRIAL: NCT00928720
Title: Cranial Electrical Stimulation Effects on Symptoms in Persons With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Ann G Taylor, Professor of Nursing, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 14203
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; pain; sleep disturbance; fatigue; depression; functional magnetic resonance imaging
MeSH Terms: conditions — Fibromyalgia; Pain; Parasomnias; Fatigue; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CES device (Active Comparator): Participants will use the device for 60 minutes each day for 8 weeks.
  Interventions: Device: CES device
- Sham device (Sham Comparator): Participants will use the device for 60 continuous minutes each day for 8 weeks. The sham device will look the same as the active CES device; however, no electrical stimulation will be present in the sham device.
  Interventions: Device: sham device
- Usual care alone (No Intervention): No intervention; participants will receive usual medical care

INTERVENTIONS:
Device: CES device — Participants will use the device for 60 continuous minutes each day for 8 weeks. The CES device will be preset at the factory to provide a maximum of 60 minutes of modified square-wave biphasic stimulation at 0.5 Hz and 100µA, the lowest setting that has been used in previous studies with patients with FM.
  Other Names: Alpha-Stim
  Arms: CES device
Device: sham device — The sham device will look the same as the active CES (Alpha-Stim); however, no electrical stimulation will be present in the sham device.
  Arms: Sham device

SUMMARY:
The purpose of this study is to determine the effects of mild cranial electrical stimulation on pain, fatigue, sleep disturbances, perceived stress, blood pressure, and functional status in persons with fibromyalgia.

DETAILED DESCRIPTION:
Central pain networks in the brain are dysregulated in persons with fibromyalgia (FM). Thus, the investigators propose that cranial electrical stimulation (CES) that works on the brain may ameliorate symptoms of FM by interacting with the central pain networks. The specific aims of this randomized, controlled, three-group pilot study design are to: (1) determine differences in pain over time between the active CES, sham device, and usual care (UC) groups; (2) explore differences in brain activity in pain processing regions (i.e., cingulate, insula, prefrontal and somatosensory cortices, amygdala, and thalamus) between the active CES, sham device, and UC groups in a subset of 12 participants (6 in each device group); (3) determine the effects of CES on other symptoms (fatigue, sleep disturbances, depression, perceived stress) and functional status, and blood pressure over time between the active CES, sham device, and UC groups; and (4) determine the amount of influence that selected psychological factors (negative affect, catastrophizing, and other personality characteristics) have on group differences in pain, other symptoms, functional status, and brain activity.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic criteria for FM established by the American College of Rheumatology
* have initial pain level equal to or greater than 3 on a NRS 0-10
* have stable medication use related to FM for at least 4 weeks
* be able to read, write, and understand the English language

Exclusion Criteria (all participants):

* pregnant or breastfeeding
* epilepsy or history of seizures
* presence of pacemakers and/or other implanted devices

Exclusion Criteria (subset of 12 participants who wil have fMRIs):

* conditions that would not permit an fMRI (e.g., certain types of metal or metallic objects in body, diaphragm or intrauterine device, dermal patches, ear or eye implants, implanted electrical stimulators, artificial heart valve, implanted catheter or tube, tattoos, claustrophobia; or weight more than 275 lbs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann G Taylor, EdD, RN, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for the Study of Complementary and Alternative Therapies, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CES Device: cranial electrical stimulation (CES) device (Alpha-Stim): Participants will use the device for 60 continuous minutes each day for 8 weeks. The CES device will be preset at the factory to provide a maximum of 60 minutes of modified square-wave biphasic stimulation at 0.5 Hz and 100µA, the lowest setting that has been used in previous studies with patients with FM.
- Usual Care Alone: No intervention; usual medical care for fibromyalgia
Period: Overall Study
Arm/Group | CES Device | Sham Device | Usual Care Alone
Started | 19 | 20 | 18
Completed | 17 | 14 | 15
Not Completed | 2 | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Usual Care Alone: No intervention; participants will received usual medical care for fibromyalgia
- Total: Total of all reporting groups
Arm/Group | CES Device | Sham Device | Usual Care Alone | Total
Number analyzed (Participants) | 17 | 14 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (10.6) | 51.5 (10.9) | 48.6 (9.8) | 50.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 14 | 43
  Male | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 17 | 14 | 15 | 46
Pain Numeric Rating Scale [Mean (Standard Deviation); unit: units on a scale] — A Numeric Rating Scale to capture average pain. The scales ranges from 0 (no pain) to 10 (worst pain imaginable).
  units on a scale | 5.8 (1.9) | 5.7 (1.6) | 6.0 (2.1) | 5.8 (1.8)
Fatigue [Mean (Standard Deviation); unit: units on a scale] — A Numeric Rating Scale to capture present fatigue. The scales ranges from 0 (no fatigue) to 10 (worst fatigue imaginable).
  units on a scale | 6.12 (1.89) | 6.66 (2.0) | 6.85 (1.74) | 6.53 (1.89)
Fibromyalgia impact [Mean (Standard Deviation); unit: units on a scale] — The Fibromyalgia Impact Questionnaire is a brief assessment and evaluation instrument consisting of 19 items to measure patient status, progress, and outcomes of patients with fibromyalgia over the past week. The measure is self-administered and takes approximately 5 minutes to complete. Total scores range from 0 to 80, with 0 indicating no impact and 80 indicating maximum impact, thus a higher score indicating more negative impact.
  units on a scale | 61.36 (18.2) | 65.98 (17.9) | 66.31 (16.9) | 64.51 (17.5)
Depression [Mean (Standard Deviation); unit: units on a scale] — The Center for Epidemiological Studies-Depression (CES-D) scale is a 20-item measure that asks the individual to rate how often over the past week s/he has experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item. Scores range from 0 to 60, with high scores indicating greater depressive symptoms. The CES-D also provides cutoff scores (e.g., 16 or greater) that aid in identifying individuals at risk for clinical depression.
  units on a scale | 23.9 (11.8) | 29.5 (13.7) | 24.1 (14.2) | 26.0 (13.3)
General sleep disturbance [Mean (Standard Deviation); unit: units on a scale] — The General Sleep Disturbance Scale (GSDS) is a subjective measure of sleep disturbance that contains 21 items rating the frequency of specific sleep problems during the past week from 0 to 7. Each item is rated on a numeric rating scale ranging from 0 to 7 and the total 21 items are summed to calculate total score ranging from 0 (no disturbance) to 147 (extreme disturbance); higher scores indicate greater sleep disturbances.
  units on a scale | 3.75 (0.94) | 4.01 (0.80) | 3.6 (0.86) | 3.8 (0.87)
Daily stress impact [Mean (Standard Deviation); unit: units on a scale] — The Daily Stress Inventory is a 58-item measure designed to quantify individuals' perceived daily stress by rating the stressfulness of the events identified on a Likert-type scale from 1 to 7. Three daily scores are derived for each individual: (1) number of events that are scored as having occurred (Frequency), (2) sum of the total of the impact rating of these events (Summary, and (3) average impact rating of the events (the AIR, which is obtained by dividing the Summary score by the Frequency Score). Scores range from 1 to 58, with higher scores indicating higher levels of stress.
  units on a scale | 3.86 (1.2) | 3.05 (1.1) | 3.39 (1.3) | 3.44 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Using Numeric Rating Scale
Description: A Numeric Rating Scale ranging from 0 (no pain) to 10 (worst pain imaginable) to capture present pain intensity
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Usual Care Alone: No intervention; participants will receive usual medical care for fibromyalgia
Arm/Group | CES Device | Sham Device | Usual Care Alone
Number analyzed (Participants) | 17 | 14 | 15
units on a scale | 5.12 (1.69) | 6.36 (2.11) | 6.62 (1.94)
Statistical Analysis 1: Comparison: Usual Care Alone; Test type: Superiority; p = 0.045, Mixed Models Analysis; Mean Difference (Final Values) = 0.05

2. Secondary Outcome: Fatigue Using Lee's Fatigue Scale
Description: A Numeric Rating Scale ranging from 0-10 to capture present levels of fatigue using the fatigue subscale of Lee's Fatigue Scale
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CES Device | Sham Device | Usual Care Alone
Number analyzed (Participants) | 17 | 14 | 15
units on a scale | 4.97 (2.45) | 6.38 (2.2) | 6.83 (2.35)

3. Secondary Outcome: General Sleep Disturbance Scale
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CES Device | Sham Device | Usual Care Alone
Number analyzed (Participants) | 17 | 14 | 15
units on a scale | 2.79 (1.07) | 3.86 (1.17) | 3.53 (1.14)

4. Secondary Outcome: Depression Using the CES-D
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CES Device | Sham Device | Usual Care Alone
Number analyzed (Participants) | 17 | 14 | 15
units on a scale | 16.5 (10.1) | 28.63 (14.9) | 23.42 (13.2)

5. Secondary Outcome: Perceived Stress Using Numeric Rating Scale
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CES Device | Sham Device | Usual Care Alone
Number analyzed (Participants) | 17 | 14 | 15
units on a scale | 3.93 (2.4) | 5.64 (2.66) | 5.29 (2.61)

6. Secondary Outcome: Functional Status Using the Fibromyalgia Index Questionnaire
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CES Device | Sham Device | Usual Care Alone
Number analyzed (Participants) | 17 | 14 | 15
units on a scale | 45.05 (16.3) | 70.1 (22.3) | 63.2 (19.9)

ADVERSE EVENTS:
Arm/Group | CES Device | Sham Device | Usual Care Alone
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No